CLINICAL TRIAL: NCT02795793
Title: A Prospective Randomised Controlled Non-inferiority Study to Evaluate the Effectiveness and Safety (APRES) of Non-operative Management in Children With Acute Uncomplicated Appendicitis
Brief Title: Non-operative Management for Appendicitis in Children
Acronym: APRES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sydney Children's Hospitals Network (Other)
Responsible Party: Principal Investigator, Dr Susan Adams, Dr Susan Adams, Sydney Children's Hospitals Network
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HERC/15/SCHN/266
Record Dates: First submitted 2016-05-29; First posted 2016-06-10 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Acute Focal Appendicitis; Appendicitis
Keywords: appendicitis; non-operative management; children; pediatric
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non-operative management group (NOM) (Experimental): Children in the NOM group will receive intravenous Piperacillin with Tazobactam (Tazocin) 100mg/kg/dose every 8 hours for at least 24 hours, and they will be observed and reassessed within 24 hours after randomisation. A further 24 hours of intravenous Piperacillin with Tazobactam therapy will be offered to children in invariable condition. A clinical decision will be made by the attending surgeon to offer OM if a patient's condition deteriorates at any time, or if a patient has failed to improve after 48 hours of intravenous antibiotic therapy. Once the patient is clinically improving and tolerating oral intake, the antibiotic regimen will be changed to oral Amoxicillin plus Clavulanic acid (Augmentin) 22.5mg/kg/dose twice per day to complete a total seven day course of antibiotics. Oral Ciprofloxacin 15mg/kg/dose twice daily and oral Metronidazole 10mg/kg/dose twice daily will be offered to children who are known to have an intolerance or allergy to Amoxicillin or Clavulanic acid.
  Interventions: Drug: Non-operative management group (NOM)
- Appendectomy group (Operative management, OM) (Active Comparator): Children allocated to OM may receive preoperative antibiotic prophylaxis as clinically indicated. Appendicectomy will be performed laparoscopically, or via open surgery according to the surgeon's standard practice. Postoperative antibiotic treatment will be determined on the basis of intraoperative findings in accordance with the institutional practice. The appendix specimen will be examined by a paediatric pathologist, and the formal histopathology report will be recorded.
  Interventions: Procedure: Appendectomy group (Operative management, OM)

INTERVENTIONS:
Drug: Non-operative management group (NOM) — With intravenous Piperacillin with Tazobactam (Tazocin)
  Arms: Non-operative management group (NOM)
Procedure: Appendectomy group (Operative management, OM)
  Arms: Appendectomy group (Operative management, OM)

SUMMARY:
This study is designed to determine the safety and efficacy of non-operative antibiotic management of clinically diagnosed acute uncomplicated appendicitis in children. Enrolled patients will be randomised and an allocation ratio of 1:1 will be made via weighted minimisation, where half of the patients will receive non-operative management with intravenous Piperacillin with Tazobactam, while the other half will have an appendicectomy.

DETAILED DESCRIPTION:
Appendicectomy for acute appendicitis is one of the most commonly performed paediatric emergency operations in Australia. This standard treatment of acute uncomplicated appendicitis (AUA) has remained largely unchallenged since its introduction in the late nineteenth century, under the assumption that AUA progresses to perforation and thus complications should an operation be withheld. However, appendicectomy via laparoscopic or open approach is not without its risks.

Non-operative management (NOM) with antibiotics has been increasingly accepted as mainstay therapy for many intra-abdominal infections. In fact, children with appendicitis complicated by perforation, abscess or phlegmon formation are often preferentially treated non-operatively with antibiotic therapy, with or without percutaneous drainage. Systematic reviews and meta-analyses have demonstrated that antibiotics are a safe and effective treatment for AUA in adults and there is growing evidence that NOM is safe and effective in children.

Primary objectives:

To determine the safety and efficacy of non-operative antibiotic management of clinically diagnosed likely AUA in children.

Secondary objectives:

1. To compare the safety and efficacy of NOM of clinically diagnosed likely AUA with operative management (OM) in children.
2. To assess the cost-effectiveness of NOM of clinically diagnosed likely AUA against OM in children.
3. To assess the feasibility and acceptability of NOM of appendicitis in children.

This study will enrol 226 patients, age 5-16 years, with acute uncomplicated appendicitis at two tertiary children's hospitals. Allocation ratio of 1:1 will be made via weighted minimisation using the following criteria: age (5-8 years or 9-16 years), gender (male or female), and duration of symptoms (<48 or >48 hours).

ELIGIBILITY:
Inclusion Criteria:

1. Age between 5 and 15 years;
2. Clinical diagnosis by at least one paediatric surgeon (or duty surgical registrar) of acute uncomplicated appendicitis based on with a combination of clinical, laboratory and/or imaging findings; that before the study would have led to the decision to recommend been subjected to an appendicectomy.

Exclusion Criteria: if one or more of the following is assessed to be present

1. Suspicion of perforated appendicitis on the basis of generalised peritonitis and/or imaging studyA diagnosis of perforated or complicated appendicitis (e.g. peritonitis, appendiceal mass) is made on the basis of clinical, laboratory and/or imaging findings;
2. Previous non-operative treatment of acute appendicitis;
3. Age younger than 5 years or older than 16 years;
4. Known intolerance or allergy to Piperacillin with Tazobactam;
5. Known history of inflammatory bowel disease, or other chronic abdominal pain syndrome;
6. Known concurrent significant illness;
7. Unable to obtain informed consent from parents or guardian;
8. Known to have a cognitive impairment, an intellectual disability or a mental illness that would impair participation.

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 226 (Estimated)
Dates: Start 2016-05; Primary Completion 2019-05 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Unplanned or unnecessary operation(s) and complications | 30 days

SECONDARY OUTCOMES:
Unplanned or unnecessary operation, or complications | 6 months
Length of primary hospital stay | 72 hours
  Time of randomisation to discharge
Treatment-related complications | 12 months
Redamission and Emergency Department presentation | 12 months
Cost of treatment in Australian Dollars (AUD) | 12 months
Return to school from time of randomisation | 30 days
Return to normal activities from time of randomisation | 30 days

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales

REFERENCES:
- [Derived] Xu J, Liu YC, Adams S, Karpelowsky J. Acute uncomplicated appendicitis study: rationale and protocol for a multicentre, prospective randomised controlled non-inferiority study to evaluate the safety and effectiveness of non-operative management in children with acute uncomplicated appendicitis. BMJ Open. 2016 Dec 21;6(12):e013299. doi: 10.1136/bmjopen-2016-013299. PMID 28003294